CLINICAL TRIAL: NCT00106353
Title: A Phase I/II Safety and Exploratory Pharmacogenomic/Pharmacodynamic Study of Intravenous Temsirolimus (CCI-779) in Pediatric Subjects With Relapsed/Refractory Solid Tumors
Brief Title: Study Evaluating Biomarkers In Relapsed/Refractory Pediatric Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3066K1-139
Record Dates: First submitted 2005-03-22; First posted 2005-03-23 (Estimated); Results first posted 2011-01-11 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma; Neoplasms
Keywords: Pediatric Tumors
MeSH Terms: conditions — Adenocarcinoma; Neoplasms | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1.0 (Experimental)
  Interventions: Drug: Torisel

INTERVENTIONS:
Drug: Torisel — 60-minute intravenous (IV) infusion once weekly to pediatric subjects with advanced solid tumors. Part 1 is an ascending-dose study to evaluate the safety of IV temsirolimus given once weekly to subjects ages 1 to 21 years with advanced solid tumors disease that is recurrent or refractory to standard therapy or for whom standard therapy is not available. (enrollment completed) Part 2 will be conducted in three groups of children with refractory or relapsed pediatric solid tumors. Subjects with the following tumor types will be enrolled: neuroblastoma, rhabdomyosarcoma, and high-grade gliomas. Subjects will receive IV temsirolimus once weekly until disease progression or unacceptable toxicity.
  Other Names: temsirolimus

SUMMARY:
This is an open label, two-part study of temsirolimus given as a 60-minute intravenous (IV) infusion once weekly to pediatric subjects with advanced solid tumors.

Part 1 is an ascending-dose study to evaluate the safety of IV temsirolimus given once weekly to subjects ages 1 to 21 years with advanced solid tumors disease that is recurrent or refractory to standard therapy or for whom standard therapy is not available. (enrollment completed) Part 2 will be conducted in three groups of children with refractory or relapsed pediatric solid tumors. Subjects with the following tumor types will be enrolled: neuroblastoma, rhabdomyosarcoma, and high-grade gliomas. Subjects will receive IV temsirolimus once weekly until disease progression or unacceptable toxicity. (recruiting)

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

Part 1 only:

- Subjects with a histological diagnosis of advanced cancer (solid tumors or central nervous system [CNS] tumors) with disease that is recurrent or refractory to standard therapy or for whom standard therapy is not available (histological confirmation waived for brain stem gliomas and optic pathway tumors)

Part 2 only:

* Subjects with histologically confirmed diagnosis of refractory or relapsed: Neuroblastoma, High-grade gliomas: glioblastoma multiforme, anaplastic astrocytomas, and other high-grade gliomas (histological confirmation waived for brain stem gliomas), Rhabdomyosarcoma.
* Measurable disease (for subjects with neuroblastoma, evaluable disease as determined by a positive metaiodobenzylguanidine (MIBG) scan will also be permitted).

Exclusion Criteria:

Exclusion Criteria:

* Subjects receiving enzyme-inducing anticonvulsants.
* Pulmonary hypertension or pneumonitis
* Active infection or serious intercurrent illness
* Other exclusions apply

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2005-03; Primary Completion 2009-10 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- United States (11):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Seattle, Washington
- Canada (6):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
- France (2):
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Villejuif
- Pfizer Investigational Site, Münster, Germany
- Pfizer Investigational Site, Mexico City, Mexico City, Mexico
- Poland (2):
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Warsaw
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg

REFERENCES:
- [Derived] Geoerger B, Kieran MW, Grupp S, Perek D, Clancy J, Krygowski M, Ananthakrishnan R, Boni JP, Berkenblit A, Spunt SL. Phase II trial of temsirolimus in children with high-grade glioma, neuroblastoma and rhabdomyosarcoma. Eur J Cancer. 2012 Jan;48(2):253-62. doi: 10.1016/j.ejca.2011.09.021. Epub 2011 Oct 25. PMID 22033322

RESULTS

PARTICIPANT FLOW:
Groups:
- Temsirolimus 10 mg/m^2: Part 1: Temsirolimus 10 milligram per square meter (mg/m^2) administered intravenously once weekly over 60 minutes infusion.
- Temsirolimus 25 mg/m^2: Part 1: Temsirolimus 25 mg/m^2 administered intravenously once weekly over 60 minutes infusion.
- Temsirolimus 75 mg/m^2: Part 1: Temsirolimus 75 mg/m^2 administered intravenously once weekly over 60 minutes infusion.
- Temsirolimus 150 mg/m^2: Part 1: Temsirolimus 150 mg/m^2 administered intravenously once weekly over 60 minutes infusion.
- High-grade Glioma: Part 2: Participants with high-grade glioma were administered temsirolimus 75 mg/m^2 intravenously once weekly over 60 minutes infusion.
- Neuroblastoma: Part 2: Participants with neuroblastoma were administered temsirolimus 75 mg/m^2 intravenously once weekly over 60 minutes infusion.
- Rhabdomyosarcoma: Part 2: Participants with rhabdomyosarcoma were administered temsirolimus 75 mg/m^2 intravenously once weekly over 60 minutes infusion.
Period: Part 1
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1 | High-grade Glioma: Part 2 | Neuroblastoma: Part 2 | Rhabdomyosarcoma: Part 2
Started | 4 | 5 | 3 | 7 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 5 | 3 | 7 | 0 | 0 | 0
Not completed — Disease progression | 3 | 4 | 1 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Symptomatic deterioration | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Entered follow-up phase | 1 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Part 2
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1 | High-grade Glioma: Part 2 | Neuroblastoma: Part 2 | Rhabdomyosarcoma: Part 2
Started | 0 | 0 | 0 | 0 | 17 | 19 | 16
Completed | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 16 | 18 | 16
Not completed — Disease progression | 0 | 0 | 0 | 0 | 8 | 14 | 13
Not completed — Death | 0 | 0 | 0 | 0 | 3 | 0 | 1
Not completed — Symptomatic deterioration | 0 | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Participants received temsirolimus intravenously once weekly over 60 minutes infusion in dose escalation schemes of 10 mg/m^2, 25 mg/m^2, 75 mg/m^2 and 150 mg/m^2.
- Part 2: Participants with high-grade glioma, neuroblastoma and rhabdomyosarcoma were administered temsirolimus 75 mg/m^2 intravenously once weekly over 60 minutes infusion.
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2 | Total
Number analyzed (Participants) | 19 | 52 | 71
Age, Customized [Number; unit: participants]
  Greater than or equal to(>=)1 to less than16 years | 12 | 42 | 54
  >=16 to less than 18 years | 2 | 3 | 5
  >=18 to less than or equal to 21 years | 5 | 7 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 17 | 25
  Male | 11 | 35 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs): Part 1
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to End of Treatment (EOT) (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- Temsirolimus 10 mg/m^2: Part 1: Temsirolimus 10 milligrams per square meter (mg/m^2) administered intravenously once weekly over 60 minutes infusion.
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 5 | 3 | 7
participants
  AEs | 4 | 5 | 3 | 7
  SAEs | 2 | 2 | 2 | 3

2. Secondary Outcome: Number of Participants Who Reached Maximum Tolerated Dose Due to Dose Limiting Toxicity: Part 1
Description: Maximum tolerated dose (MTD) defined as the dose level at which >=2 of 3 participants or >=2 of 6 participants if the dose level had been expanded, experienced a dose limiting toxicity (DLT) by day 21 after the first dose of study treatment. DLT defined as failure to recover to NCI-CTCAE version 3.0 grade 0 to 2 (or within 1 grade of starting values for pre-existing laboratory abnormalities) from a treatment-related toxicity within 3 weeks (leading to a treatment delay of > 3 weeks) unless the investigator and the medical monitor agree that the subject should remain in the study.
Time Frame: Baseline up to Month 6
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 5 | 3 | 7
participants | 0 [9.40 to 10.11] | 0 [23.20 to 25.40] | 0 [71.77 to 75.26] | 2 [89.21 to 156.50]

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax): Part 1
Time Frame: 0 (pre-dose), 1, 2, 6, 24, and 168 hours (hrs) post-dose of Cycle 1 and 0 (pre-dose), 1, 2, 6, 24, 72, 96, and 168 hrs post-dose of Cycle 2 (cycles are approximately 21 days)
Population: Safety population included all participants who received at least 1 dose of study medication. Here, 'n' signifies those participants who were evaluable for particular cycle for each group respectively.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 5 | 3 | 7
nanogram per milliliter (ng/mL)
  Cycle 1 (n = 4, 5, 3, 7) | 307 (91.3) | 487 (141) | 480 (135) | 9230 (18200)
  Cycle 2 (n = 4, 4, 3, 5) | 252 (98.3) | 403 (128) | 807 (279) | 2570 (1110)

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax): Part 1
Time Frame: 0 (pre-dose), 1, 2, 6, 24, and 168 hrs post-dose of Cycle 1 and 0 (pre-dose), 1, 2, 6, 24, 72, 96, and 168 hrs post-dose of Cycle 2 (cycles are approximately 21 days)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 5 | 3 | 7
hr
  Cycle 1 (n = 4, 5, 3, 7) | 1 (0.143) | 1.1 (0.074) | 1.3 (0.231) | 1.1 (0.218)
  Cycle 2 (n = 4, 4, 3, 5) | 1.1 (0.236) | 1.7 (0.983) | 1.2 (0.202) | 1.2 (0.212)

5. Secondary Outcome: Plasma Decay Half-Life (t1/2): Part 1
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 4
Population: Safety population included all participants who received at least 1 dose of study medication. Here, the 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure for each group respectively. Here, 'n' signifies those participants who were evaluable for particular cycle for each group respectively.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 4 | 3 | 5
hr
  Cycle 1 (n = 4, 4, 1, 4) | 10.6 (0.556) | 16.4 (6.9) | 24 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 19.3 (10.5)
  Cycle 2 (n = 4, 3, 3, 5) | 14.4 (4.42) | 14.3 (10.4) | 25.4 (1.83) | 24.2 (7.58)

6. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)]: Part 1
Description: AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t).
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 5 | 3 | 7
hr*ng/mL
  Cycle 1 (n = 4, 5, 3, 7) | 1670 (730) | 3890 (3190) | 3750 (2420) | 9680 (12800)
  Cycle 2 (n = 4, 4, 3, 5) | 1520 (583) | 1930 (1090) | 3420 (1230) | 4850 (1810)

7. Secondary Outcome: Area Under the Concentration-Time Curve (AUC): Part 1
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 4 | 3 | 5
hr*ng/mL
  Cycle 1 (n = 4, 4, 1, 4) | 2000 (959) | 4640 (3430) | 2810 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 13000 (17000)
  Cycle 2 (n = 4, 3, 3, 5) | 1600 (540) | 2580 (768) | 3500 (1140) | 4960 (2000)

8. Secondary Outcome: Clearance (CL): Part 1
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liter/hr
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 4 | 3 | 5
Liter/hr
  Cycle 1 (n = 4, 4, 1, 4) | 7.02 (3.68) | 10.4 (6.45) | 38.1 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 47.9 (45.8)
  Cycle 2 (n = 4, 3, 3, 5) | 8.99 (5.27) | 13.8 (9.06) | 30.6 (15.5) | 39 (24.4)

9. Secondary Outcome: Volume of Distribution at Steady State (Vss): Part 1
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 4 | 3 | 5
Liter
  Cycle 1 (n = 4, 4, 1, 4) | 85.2 (35) | 189 (44.2) | 783 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 512 (689)
  Cycle 2 (n = 4, 3, 3, 5) | 250 (290) | 201 (132) | 601 (347) | 353 (130)

10. Secondary Outcome: Percentage of Participants With Best Overall Response: Part 1
Description: Best overall response is the best response recorded from baseline until disease progression or recurrence. Measured as CR, PR, SD, PD, or Unknown. CR=disappearance of all primary and metastatic lesions. PR=at least a 50% decrease in primary disease measurement. SD=no new lesions; decrease of <50% in all lesions with no lesion increasing >25%. PD=any new lesion; at least a 25% increase in any disease measurement (reference smallest disease measurement recorded since start of treatment); or appearance of 1 or more new lesions. Tumor response considered Unknown if assessment prior to Day 37.
Time Frame: Baseline until disease progression or recurrence (actual greatest response day is up to Day 49)
Population: Efficacy evaluable population included all participants who received at least 3 doses of study medication. Here, the 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure for each group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 4 | 3 | 7
percentage of participants
  Complete response | 1 | 0 | 0 | 0
  Partial response | 0 | 0 | 0 | 0
  Stable disease | 0 | 2 | 3 | 2
  Progressive disease | 3 | 2 | 0 | 3
  Unknown response | 0 | 0 | 0 | 2

11. Secondary Outcome: Percentage of Participants Exhibiting Freedom From Progression at Week 12: Part 2
Description: Freedom from progression measured as Stable Disease (SD) or better and no Progressive Disease (PD); (CR+VGPR+Mixed Response [MR]+PR+SD). CR=disappearance of all primary and metastatic lesions. VGPR=disappearance of all metastatic lesions. MR=no new lesions; at least 50% decrease in any 1 disease measurement with <50% decrease in any other disease measurement or an increase of <25% in any lesion). SD=no new lesions; decrease of <50% in all lesions with no lesion increasing >25%. PD=at least a 25% increase in any disease measurement; or the appearance of 1 or more new lesions.
Time Frame: Week 12
Population: Efficacy evaluable population included all participants who received at least 3 doses of study treatment. Here, the 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure for each group respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-grade Glioma: Part 2 | Neuroblastoma: Part 2 | Rhabdomyosarcoma: Part 2
Number analyzed (Participants) | 15 | 15 | 12
percentage of participants | 46.67 [21.27 to 73.41] | 40.00 [16.34 to 67.71] | 8.33 [0.21 to 38.48]

12. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs): Part 2
Description: as for outcome 1
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | High-grade Glioma: Part 2 | Neuroblastoma: Part 2 | Rhabdomyosarcoma: Part 2
Number analyzed (Participants) | 17 | 19 | 16
participants
  AEs | 17 | 19 | 16
  SAEs | 10 | 6 | 6

13. Secondary Outcome: Number of Participants With Drug Related Treatment Emergent Adverse Events (TEAEs): Part 2
Description: Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | High-grade Glioma: Part 2 | Neuroblastoma: Part 2 | Rhabdomyosarcoma: Part 2
Number analyzed (Participants) | 17 | 19 | 16
participants | 17 | 18 | 13

14. Secondary Outcome: Number of Participants With Drug Related Grade 3 and Higher Treatment Emergent Adverse Events (TEAEs): Part 2
Description: Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. NCI-CTC provides descriptive terminology for adverse event reporting. A grading (severity) scale is provided for each adverse event term. Grades range from 0 (none) to 5 (death).
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | High-grade Glioma: Part 2 | Neuroblastoma: Part 2 | Rhabdomyosarcoma: Part 2
Number analyzed (Participants) | 17 | 19 | 16
participants | 5 | 11 | 6

15. Secondary Outcome: Number of Participants Who Died: Part 2
Description: Deaths were reported from baseline throughout the 30 day period after last study treatment. After the 30 day reporting period, only deaths believed related to study treatment were to be reported (as SAEs).
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | High-grade Glioma: Part 2 | Neuroblastoma: Part 2 | Rhabdomyosarcoma: Part 2
Number analyzed (Participants) | 17 | 19 | 16
participants
  Died=Yes | 5 | 2 | 4
  Died within 30 days of last dose | 3 | 0 | 3

16. Secondary Outcome: Number of Participants With Drug Related Serious Adverse Events (SAEs): Part 2
Description: An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Participants with documented study treatment toxicity were followed weekly until recovering. After the 30 day reporting period, only SAEs believed to be related to study treatment were to be reported.
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | High-grade Glioma: Part 2 | Neuroblastoma: Part 2 | Rhabdomyosarcoma: Part 2
Number analyzed (Participants) | 17 | 19 | 16
participants | 2 | 3 | 3

17. Secondary Outcome: Number of Participants With Adverse Events Causing Temporary Stop of Study Treatment: Part 2
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Temporary interruption of study treatment may be followed by resumption of study treatment at current dose or dose modification as determined by the investigator and medical monitor.
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | High-grade Glioma: Part 2 | Neuroblastoma: Part 2 | Rhabdomyosarcoma: Part 2
Number analyzed (Participants) | 17 | 19 | 16
participants | 9 | 12 | 6

18. Secondary Outcome: Number of Participants With Adverse Events Causing Dose Reduction of Study Treatment: Part 2
Description: Dose reduction for individual participant allowed if a DLT occurred; may continue treatment following reduction by 1 to 2 dose levels (determined by investigator and medical monitor). DLT= failure to recover to National Cancer Institute Common Terminology Criteria for AEs (NCI-CTCAE) version 3.0 grade 0 to 2 (or within 1 grade of starting values for pre-existing laboratory abnormalities) from a treatment-related toxicity within 3 weeks (leading to a treatment delay of >3 weeks) unless investigator and medical monitor agree participant should remain in the study.
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | High-grade Glioma: Part 2 | Neuroblastoma: Part 2 | Rhabdomyosarcoma: Part 2
Number analyzed (Participants) | 17 | 19 | 16
participants | 5 | 10 | 6

19. Primary Outcome: Number of Participants With Drug Related Treatment Emergent Adverse Events (TEAEs): Part 1
Description: TEAEs are events that occurred on or after initial treatment that were absent before treatment or worsened during the treatment period relative to the pretreatment state. AEs that occurred within 30 days of the last administration of study treatment can be attributed to the treatment period.
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- Temsirolimus 150 mg/m^2: Part 1: Temsirolimus 150 mg/m^2 intravenously administered once weekly over 60 minutes infusion.
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 5 | 3 | 7
participants | 4 | 5 | 3 | 7

20. Primary Outcome: Number of Participants With Drug Related Grade 3 and Higher Treatment Emergent Adverse Events (TEAEs): Part 1
Description: TEAEs are events that occurred on or after initial treatment that were absent before treatment or worsened during the treatment period relative to the pretreatment state. AEs that occurred within 30 days of the last administration of study treatment can be attributed to the treatment period. National Cancer Institute (NCI)-graded Common Toxicity Criteria (CTC) provides descriptive terminology for adverse event reporting. A grading (severity) scale is provided for each adverse event term. Grades range from 0 (none) to 5 (death).
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 5 | 3 | 7
participants | 1 | 2 | 2 | 4

21. Primary Outcome: Number of Participants Who Died: Part 1
Description: as for outcome 15
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 5 | 3 | 7
participants
  Died=Yes | 3 | 1 | 0 | 0
  Died within 30 days of last dose | 2 | 0 | 0 | 0

22. Primary Outcome: Number of Participants With Drug Related Serious Adverse Events (SAEs): Part 1
Description: SAEs include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability / incapacity or are a congenital anomaly or birth defect in the offspring of a study subject. Participants with documented study treatment toxicity were followed weekly until recovering. After the 30 day reporting period, only SAEs believed to be related to study treatment were to be reported.
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 5 | 3 | 7
participants | 0 | 0 | 0 | 1

23. Primary Outcome: Number of Participants With Adverse Events Causing Temporary Stop of Study Treatment: Part 1
Description: Temporary interruption of study treatment; may be followed by resumption of study treatment at current dose or dose modification as determined by the investigator and medical monitor.
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 5 | 3 | 7
participants | 0 | 2 | 1 | 2

24. Primary Outcome: Number of Participants With Adverse Events Causing Dose Reduction of Study Treatment: Part 1
Description: Dose reduction for individual participant allowed if a dose limiting toxicity (DLT) occurred; may continue treatment following reduction by 1 to 2 dose levels (determined by investigator and medical monitor). DLT= failure to recover to National Cancer Institute Common Terminology Criteria for AEs (NCI-CTCAE) version 3.0 grade 0 to 2 (or within 1 grade of starting values for pre-existing laboratory abnormalities) from a treatment-related toxicity within 3 weeks (leading to a treatment delay of >3 weeks) unless investigator and medical monitor agree participant should remain in the study.
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 5 | 3 | 7
participants | 0 | 0 | 0 | 1

25. Primary Outcome: Number of Participants With Potentially Clinically Important (PCI) Changes in Vital Signs: Part 1
Description: Number of participants who met the criteria for PCI changes (based on baseline values before treatment); criteria defined as body temperature >39 degrees Celsius (C), respiratory rate >20 beats per minute (bpm), and systolic and diastolic blood pressure (BP) >200/110 millimeters of mercury (mmHg). Participants may be reported in more than 1 category.
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 5 | 3 | 7
participants
  Temperature >39 degrees C | 1 | 2 | 1 | 3
  Respiratory rate >20 bpm | 4 | 5 | 3 | 7
  Systolic/Diastolic BP >200/110 mmHg | 0 | 0 | 0 | 0

26. Secondary Outcome: Number of Participants With Potentially Clinically Important (PCI) Changes in Vital Signs: Part 2
Description: Number of participants who met the criteria for PCI changes (based on baseline values before treatment); criteria defined as body temperature >39 degrees C, respiratory rate >20 bpm, and systolic and diastolic BP >200/110 mmHg. Participants may be reported in more than 1 category.
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | High-grade Glioma: Part 2 | Neuroblastoma: Part 2 | Rhabdomyosarcoma: Part 2
Number analyzed (Participants) | 17 | 19 | 16
participants
  Temperature >39 degrees C | 0 | 0 | 0
  Respiratory rate >20 bpm | 16 | 18 | 14
  Systolic/Diastolic BP >200/110 mmHg | 1 | 0 | 0

27. Secondary Outcome: Number of Participants With Potentially Clinically Important (PCI) Values by National Cancer Institute Common Terminology Criteria (NCI-CTC) Grade for Laboratory Values: Part 2
Description: Number of participants who met the PCI criteria (grades 1 through 5) for laboratory values (hematology and serum chemistry). NCI-CTC provides descriptive terminology for adverse event reporting. A grading (severity) scale is provided with grades ranging from 0 (none), 1 (mild), 2 (moderate), 3 (severe), 4 (life-threatening or disabling), to 5 (death). Participants may be reported in more than 1 category.
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | High-grade Glioma: Part 2 | Neuroblastoma: Part 2 | Rhabdomyosarcoma: Part 2
Number analyzed (Participants) | 17 | 19 | 16
participants | 17 | 19 | 15

28. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax): Part 2
Time Frame: 0 (pre-dose), 1, 6, 24, 48, 72, 96, and 168 hrs post-dose of Cycle 2 (cycles are approximately 21 days)
Population: Safety population included all participants who received at least 1 dose of study medication. Here, the 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2
Number analyzed (Participants) | 35
ng/mL | 6280 (21000)

29. Secondary Outcome: Average Plasma Concentration (Cavg): Part 2
Time Frame: 0 (pre-dose), 1, 6, 24, 48, 72, 96, and 168 hrs post-dose of Cycle 2 (cycles are approximately 21 days)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2
Number analyzed (Participants) | 31
ng/mL | 82.8 (143)

30. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax): Part 2
Time Frame: 0 (pre-dose),1, 6, 24, 48, 72, 96, and 168 hrs post-dose of Cycle 2 (cycles are approximately 21 days)
Population: as for outcome 28
Measure: Median (Full Range); unit: hr
Arm/Group | Part 2
Number analyzed (Participants) | 35
hr | 1.00 [0.00 to 6.00]

31. Secondary Outcome: Plasma Decay Half-Life (t1/2): Part 2
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 1, 6, 24, 48, 72, 96, and 168 hrs post-dose of Cycle 2 (cycles are approximately 21 days)
Population: Safety population included all participants who received at least 1 dose of study medication. Here, the 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure for.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part 2
Number analyzed (Participants) | 26
hr | 30.65 (13.63)

32. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)]: Part 2
Description: as for outcome 6
Time Frame: 0 (pre-dose), 1, 6, 24, 48, 72, 96, and 168 hrs post-dose of Cycle 2 (cycles are approximately 21 days)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 2
Number analyzed (Participants) | 35
hr*ng/mL | 13100 (22700)

33. Primary Outcome: Number of Participants With Potentially Clinically Important (PCI) Values by National Cancer Institute Common Terminology Criteria (NCI-CTC) Grade for Laboratory Values: Part 1
Description: as for outcome 27
Time Frame: Baseline up to EOT (within 30 days of last dose)
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1
Number analyzed (Participants) | 4 | 5 | 3 | 7
participants | 4 | 5 | 3 | 7

34. Primary Outcome: Percentage of Participants With Objective Response (OR) at Week 12: Part 2
Description: Measured as Complete response (CR), Very good partial response (VGPR), or Partial response (PR) on at least 2 occasions greater than or equal to (>=) 4 weeks apart within first 12 weeks. CR=disappearance of all primary and metastatic lesions; Homovanillic acid, Vanillymandelic acid (HVA/VMA) normal; bone marrow immunocytology negative. VGPR=disappearance of all metastatic lesions (residual areas of uptake on bone permitted); 90 to 99 percent (%) decrease in primary disease measurement; HVA/VMA normal or both decreased >90%. PR=at least 50% decrease in primary and metastatic disease. Number of bone sites decreased by at least 50%.
Time Frame: Week 12
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | High-grade Glioma: Part 2 | Neuroblastoma: Part 2 | Rhabdomyosarcoma: Part 2
Number analyzed (Participants) | 15 | 15 | 12
percentage of participants | 0.00 | 6.67 | 0.00

35. Secondary Outcome: Area Under the Concentration-time Curve at Steady State (AUCss): Part 2
Description: AUCss is a measure of the serum concentration of the drug at steady state. It is used to characterize drug absorption.
Time Frame: 0 (pre-dose), 1, 6, 24, 48, 72, 96, and 168 hrs post-dose of Cycle 2 (cycles are approximately 21 days)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 2
Number analyzed (Participants) | 31
hr*ng/mL | 13900 (24100)

36. Secondary Outcome: Clearance (CL): Part 2
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: 0 (pre-dose),1, 6, 24, 48, 72, 96, and 168 hrs post-dose of Cycle 2 (cycles are approximately 21 days)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Part 2
Number analyzed (Participants) | 31
L/hr | 14.3 (14.0)

37. Secondary Outcome: Concentration in Plasma (Cp) and Concentration in Plasma at Time Zero (Cp Time 0): Part 1 and Part 2
Description: Pharmacokinetic parameters determined in whole blood; derived from the concentration-versus-time profiles using noncompartmental analysis method. Measured as nanograms per milliliter (ng/mL).
Time Frame: Part 1: 0 (pre-dose), 1, 2, 6, 24, and 168 hrs post-dose of Cycle 1 and 0 (pre-dose), 1, 2, 6, 24, 72, 96, and 168 hrs post-dose of Cycle 2; Part2: 0 (pre-dose), 1, 6, 24, 48, 72, 96, and 168 hrs post-dose of Cycle 2 (cycles are approximately 21 days)
Population: Data was not analyzed.
Arm/Group | Part 1 | Part 2
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Number of Participants for Change From Baseline in the Phosphorylation of Mammalian Target of Rapamycin (mTOR) Pathway Proteins: Part 1 and Part 2
Description: Optional bone marrow sampling for pharmacodynamic analysis of effects of study treatment. Data may not be collected for a majority of patients and was not to be summarized if collection was sparse.
Time Frame: Part 1:Baseline,1,2,6,24,168 hrs post-dose of Cycle 1;additional 0 (Pre-dose),24,72,96 hrs, Day 16 to 21 of cycle 2, EOT(within 30 days of last dose); Part 2:Baseline,Day16 to 21 in Cycle 2, at time of disease progression, EOT(within 30 days of last dose)
Population: Data was not analyzed.
Arm/Group | Part 1 | Part 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Temsirolimus 10 mg/m^2: Part 1: Temsirolimus 10 mg/m^2 administered intravenously once weekly over 60 minutes infusion.
- Temsirolimus 25 mg/m^2: Part 1: Temsirolimus 25 mg/m^2 intravenously administered once weekly over 60 minutes infusion.
- Temsirolimus 75 mg/m^2: Part 1: Temsirolimus 75 mg/m^2 intravenously administered once weekly over 60 minutes infusion.
Arm/Group | Temsirolimus 10 mg/m^2: Part 1 | Temsirolimus 25 mg/m^2: Part 1 | Temsirolimus 75 mg/m^2: Part 1 | Temsirolimus 150 mg/m^2: Part 1 | High-grade Glioma: Part 2 | Neuroblastoma: Part 2 | Rhabdomyosarcoma: Part 2
Serious Adverse Events (participants affected / at risk) | 2/4 | 2/5 | 2/3 | 3/7 | 10/17 | 6/19 | 6/16
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 3/3 | 7/7 | 17/17 | 19/19 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temsirolimus 10 mg/m^2: Part 1 (N=4) | Temsirolimus 25 mg/m^2: Part 1 (N=5) | Temsirolimus 75 mg/m^2: Part 1 (N=3) | Temsirolimus 150 mg/m^2: Part 1 (N=7) | High-grade Glioma: Part 2 (N=17) | Neuroblastoma: Part 2 (N=19) | Rhabdomyosarcoma: Part 2 (N=16)
Pain (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 — Organ System "General disorders" equivalent to COSTART "Body as a whole".
Fever (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sarcoma (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infection (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Organ System "Cardiac disorders" equivalent to COSTART "Cardiovascular system".
Shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 — Organ System "Gastrointestinal disorders" equivalent to COSTART "Digestive system".
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — Organ System "Nervous system disorders" equivalent to COSTART "Nervous system".
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paresis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — Organ System "Respiratory, thoracic, and mediastinal disorders" equivalent to COSTART "Respiratory system".
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coordination abnormal (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drooling (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temsirolimus 10 mg/m^2: Part 1 (N=4) | Temsirolimus 25 mg/m^2: Part 1 (N=5) | Temsirolimus 75 mg/m^2: Part 1 (N=3) | Temsirolimus 150 mg/m^2: Part 1 (N=7) | High-grade Glioma: Part 2 (N=17) | Neuroblastoma: Part 2 (N=19) | Rhabdomyosarcoma: Part 2 (N=16)
Pain (General disorders) | 2 | 2 | 3 | 2 | 0 | 0 | 0
Fever (General disorders) | 0 | 2 | 1 | 4 | 0 | 0 | 0
Infection (General disorders) | 1 | 1 | 2 | 3 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 4 | 0 | 0 | 0
Headache (General disorders) | 0 | 2 | 1 | 3 | 0 | 0 | 0
Abdominal pain (General disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0
Allergic reaction (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Back pain (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Face edema (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Accidental injury (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 1 | 4 | 0 | 0 | 0
Anorexia (Gastrointestinal disorders) | 2 | 0 | 1 | 6 | 0 | 0 | 0
Mucositis (Gastrointestinal disorders) | 2 | 1 | 1 | 3 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 4 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Oral moniliasis (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma glutamyl transpeptidase increased (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glycosuria (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 0 | 2 | 6 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 3 | 4 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 5 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 4 | 0 | 0 | 0
International normalised ratio increased (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ecchymosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fibrinogen increased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoproteinemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 4 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 4 | 0 | 0 | 0
Hyperlipemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 2 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 3 | 0 | 0 | 0
SGOT increased (Metabolism and nutrition disorders) | 2 | 2 | 2 | 2 | 0 | 0 | 0
Hypercholesteremia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 4 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0
SGPT increased (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Bilirubinemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Weight loss (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Creatinine increased (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral edema (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Organ System "Musculoskeletal and connective tissue disorders" equivalent to COSTART "Musculoskeletal system".
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy (Nervous system disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Depression (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hostility (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough increased (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 3 | 0 | 0 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 4 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Herpes simplex (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Application site reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Exfoliative dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 — Organ System "Ear and labyrinth disorders" equivalent to COSTART "Special senses".
Conjunctival injection (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — Organ System "Eye disorders" equivalent to COSTART "Special senses".
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lacrimation disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Local reaction to procedure (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Organ System "Investigations" equivalent to COSTART "Adverse event associated with miscellaneous factors".
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 5
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 5 | 6 | 6
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Exophthalmos (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 6 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 4
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal discharge (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 5 | 3
Tooth impacted (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 5 | 2 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Device occlusion (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 6 | 6 | 5
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 9 | 4
Ulcer (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyoderma (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 5 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Radiation injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 6 | 7 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 6 | 5
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 4 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 6 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Blood fibrinogen increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 4 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood magnesium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 3 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood pressure decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 4 | 6 | 2
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 6 | 1
High density lipoprotein decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 4 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 4 | 7 | 2
Respiratory rate (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 3
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 5 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 6 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 3
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 6 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 4 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 5 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Accessory nerve disorder (Nervous system disorders) | 0 | 0 | 0 (0) | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 4 | 4
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 4
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Urethral pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Urogenital haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 5 | 6 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1
Suffocation feeling (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail bed tenderness (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 5 | 3 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nail operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.